CLINICAL TRIAL: NCT05874921
Title: uTRACT Jelmyto Registry: A Multicenter, Prospective and Retrospective Registry to Evaluate Real World Experience and Outcomes of Patients With Upper Tract Urothelial Cancer (UTUC) Treated With Jelmyto
Brief Title: uTRACT Jelmyto Registry: A Registry of Patients With Upper Tract Urothelial Cancer (UTUC) Treated With Jelmyto
Acronym: uTRACT
Status: Recruiting | Type: Observational
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UT004
Record Dates: First submitted 2022-12-22; First posted 2023-05-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma; Urothelial Carcinoma Recurrent; Urothelial Carcinoma Ureter; Urothelial Carcinoma Ureter Recurrent; Urothelial Cancer of Renal Pelvis; Urothelial Carcinoma of the Renal Pelvis and Ureter; Carcinoma, Transitional Cell; Transitional Cell Carcinoma of Renal Pelvis
Keywords: Upper Tract Urothelial Cancer; UTUC; UGN-101; Mitomycin C; TCC; Ureteral; Upper Tract; Carcinoma; Kidney; Renal; Gel; Local; Prolonged Release; Slow Release; Kidney Sparing; Recurrence; Neoplasms by Histologic Type; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Antibiotics, Antineoplastic; Antineoplastic Agents; Alkylating Agents; Nucleic Acid Synthesis Inhibitors; Enzyme Inhibitors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma; Recurrence; Neoplasms by Histologic Type; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site | interventions — Mitomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Jelmyto: Patients with UTUC treated with Jelmyto
  Interventions: Drug: Jelmyto (mitomycin) for pyelocalyceal solution

INTERVENTIONS:
Drug: Jelmyto (mitomycin) for pyelocalyceal solution — The dose of Jelmyto to be instilled is 4 mg per mL via ureteral catheter or a nephrostomy tube, with total instillation volume based on volumetric measurements using pyelography, not to exceed 15 mL (60 mg of mitomycin).
  Instill Jelmyto once weekly for six weeks. For patients with a complete response 3 months after Jelmyto initiation, Jelmyto instillations may be administered once a month for a maximum of 11 additional instillations.
  Other Names: Jelmyto; UGN-101

SUMMARY:
The purpose of this registry is to evaluate real world experience and outcomes of patients with Upper Tract Urothelial Cancer (UTUC) treated with Jelmyto in the United States.

DETAILED DESCRIPTION:
Patients may be enrolled prospectively, at the time of receiving Jelmyto, or after receiving Jelmyto for retrospective data capture and prospective follow up. Patients will be followed until 3 years after the first dose of Jelmyto or death.

Data will be captured to address specific clinical questions and data gaps related to real world use of Jelmyto.

Example clinical questions:

1. How is Jelmyto used in the real world setting?
2. What adverse events (AEs) and at what rates and time points are they observed in the real world setting?
3. What is the disease volume before and after resection/ablation prior to treating with Jelmyto?
4. Did the use of Jelmyto impact clinical decision making and management?
5. What is the complete response (CR) rate, duration of response, and rate of progression, including subgroups of interest?
6. What are the rates of, time to, and pathology at radical nephroureterectomy (RNU) by response to treatment and number of Jelmyto doses received?
7. What are outcomes for non-responders or partial responders? What are the rates of surgical and therapeutic treatment options received following response assessment, including additional Jelmyto?
8. What was the outcome of patients with solitary kidney and/or chronic kidney disease (CKD)? Did Jelmyto prevent dialysis by avoiding nephrectomy in solitary kidney or in patients with baseline CKD?
9. What is the rate and timing of bladder cancer occurrence and/or recurrences?

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old and capable of giving informed consent.
* Diagnosis of UTUC.
* Receipt of at least 1 dose of JELMYTO after FDA approval (15 Apr 2020).

Exclusion Criteria:

* Incapable of giving informed consent (e.g., incarcerated individuals, individuals with dementia).
* Receipt of 1 or more doses of JELMYTO (also referred to as UGN-101 or Mitogel in clinical development) before FDA approval (on or before 15 Apr 2020).
* Pregnancy or lactation.
* Unable to comply with protocol requirements (for prospective data capture).
* Any medical or mental condition(s) that makes participation in the Registry inadvisable in the opinion of the Investigator (for prospective data capture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with UTUC who have been treated, are currently undergoing treatment, or will be treated with JELMYTO.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Rate of CR or no evidence of disease (NED) at first evaluation post-treatment | 3 months

SECONDARY OUTCOMES:
Duration of response | 3 years
Rate of progression | 3 years
Rates and clinical significance of AEs | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — UT Southwestern Medical Center at Dallas; Adam Feldman, MD, Principal Investigator — Massachusett's General Hospital; Solomon Woldu, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (22):
- United States (22):
  - Providence St. Johns Health Center, Santa Monica, California
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center of Florida, Inc., Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Inc., Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - The State University of Iowa, Iowa City, Iowa
  - Chesapeake Urology, Baltimore, Maryland
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Mass General Hospital (MGH), Boston, Massachusetts
  - The Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Missouri, Columbia, Missouri
  - Rutgers, New Brunswick, New Jersey
  - The Feinstein Institutes for Medical Research, Lake Success, New York
  - NYU Grossman School of Medicine, New York, New York
  - SUNY Upstate, Syracuse, New York
  - The University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas